CLINICAL TRIAL: NCT07133529
Title: Decision-making and Food Intake ("Buffet Study")
Brief Title: Decision-making and Food Intake
Acronym: Buffet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Responsible Party: Principal Investigator, Prof. Dr. Soyoung Q Park, Prof. Dr., German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Buffet
Record Dates: First submitted 2025-07-29; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Behavior; Hormones; Stress; Cognition; Food Intake
Keywords: Decision-making; Food intake; Food uncertainty
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perceived food uncertainty (Experimental)
  Interventions: Behavioral: Perceived food uncertainty
- Perceived food certainty (Experimental)
  Interventions: Behavioral: Perceived food certainty

INTERVENTIONS:
Behavioral: Perceived food uncertainty — Participants remain unaware of both the scheduled time and the length of the next meal.
  Arms: Perceived food uncertainty
Behavioral: Perceived food certainty — Participants are aware of both the scheduled time and the length of the next meal.
  Arms: Perceived food certainty

SUMMARY:
The study will investigate how the expectation of food availability impacts the response to food cues, mood, interoceptive awareness, and consumption of food intake in healthy, naturally cycling women.

DETAILED DESCRIPTION:
In this within-subjects, randomized crossover study, we will probe how perceived meal availability shapes eating behavior, cognition, and metabolic markers in healthy, naturally cycling women. Each woman attends two appointments in the afternoon (starting at 12 pm after an overnight fast): one in which meal timing and duration are fully disclosed ("certain" condition) and one in which that information is intentionally withheld ("uncertain" condition). During each appointment, participants first undergo a set of cognitive and behavioral tests, then are invited to sample ad libitum from a 30-item buffet under the respective certainty or uncertainty instructions. Venous blood is collected at six fixed intervals to measure fluctuations in ghrelin, leptin, insulin, glucose, and cortisol. To capture real-world eating patterns, participants also log all intake in a smartphone food-tracking app for three days leading up to the initial session.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women (age: 18-35 years) with a regular menstrual cycle (25-32 days)
* Legally competent/Consent to participate
* Language proficiency in German (native speaker, fluent)
* Physically and mentally healthy
* Body mass index (BMI) of 18.5 - 30 kg/m2

Exclusion Criteria:

* Current or use of hormonal contraceptives in the previous 6 months
* Current use of hormonal intra-uterine devices (IUDs)
* Previous or current pregnancy
* Diagnosed psychological or metabolic disorder
* Former or current illnesses of:

  1. Brain or mind (including anxiety disorders, depression, eating disorders, personality disorders, alcohol, drugs or drug or non-substance dependence, neurological disorders other than occasional headache, psychiatric or neurological abnomalities)
  2. Heart or blood circulation/cardiovascular disease (myocardial infarction, stroke, hypertension, hypotension, having a pacemaker)
  3. Gastro-intestinal disorders (e.g. colon diseases, irritable bowel syndrome, Crohn's disease)
  4. Endocrine disorders (e.g. thyroid disorders)
  5. Other serious past or present medical conditions (for example, metabolic syndrome, diabetes)
* Other serious health problems or current severe mental or physical stress.
* Blood clotting disorder
* Fear of drawing blood
* Severe anemia
* Previously diagnosed hypoglycemia episodes
* Regular intake of medication (e.g. Antidepressant/anti-anxiety medication)
* Blood donation within 4 weeks before the study appointment
* Intake of anticoagulant medications
* illegal drug consumption
* smoking or nicotine consumption
* extreme athletes
* vegetarians or vegans or any other dietary restrictions due to allergies or intolerances
* shift workers

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Laboratory food intake | On 1st and 2nd visit (after approximately 30 days)
  Food consumed during a laboratory ad libitum buffet task, in which participants are able to order and consume different foods from a menu of their own liking.
Food-specific inhibitory control | On 1st and 2nd visit (after approximately 30 days)
  Food-specific inhibitory control measured by a go/no-go task adapted from Teslovich et al., 2014.
Risk propensity on a decision-making task | On 1st and 2nd visit (after approximately 30 days)
  In this task, participants decide between a risky/gamble or safe option, based on a paradigm by Liu et al., 2021.
Delay Discounting behavior in a computerized task | On 1st and 2nd visit (after approximately 30 days)
  In this task, participants are asked to choose between an immediate and delayed monetary reward, based on a task paradigm by Eisenstein et al., 2015.
Range adaptation in reinforcement learning | On 1st and 2nd visit (after approximately 30 days)
  Range adaptation in the context of a reinforcement learning task is assessed using a paradigm described by Gueguen et al., 2024.
Behavioral economic paradigm | On 1st and 2nd visit (after approximately 30 days)
  In this task, participants manage a shared resource by deciding how much to extract from a common pool over multiple rounds. Based on their individual extraction, participants receive a monetary reward, which is reduced once the group exceeds a predefined extraction limit. Adapted from Lagenbach et al., 2019.
Heart rate | On 1st and 2nd visit (after approximately 30 days)
  Resting-state and task-based heart rate, measured with a three-point electrocardiogram (ECG)
Heart-rate variability | On 1st and 2nd visit (after approximately 30 days)
  Resting-state and task-based heart-rate variability measured with a three-point electrocardiogram (ECG). Respiratory activity will also be recorded using a breathing belt to correct for breathing-related artifacts.
Electrodermal activity | On 1st and 2nd visit (after approximately 30 days)
  Resting-state and task-based skin conductance measured with two electrodermal activity electrodes placed on the fingers of the non-dominant hand.
Subjective stress levels | On 1st and 2nd visit (after approximately 30 days)
  Subjective stress levels are measured on a semi-continous scale from 1 (not at all) to 100 (extremely) repeatedly during each visit to assess stress responses to perceived food availability. Higher scores indicate greater stress.
Subjective hunger levels | On 1st and 2nd visit (after approximately 30 days)
  Subjective hunger levels are measured on a semi-continous scale from 1 (not at all) to 100 (extremely) repeatedly during each visit to assess changes in subjective hunger ratings in response to perceived food availability. Higher scores indicate greater hunger.
Subjective fullness levels | On 1st and 2nd visit (after approximately 30 days)
  Subjective fullness levels are measured on a semi-continous scale from 1 (not at all) to 100 (extremely) repeatedly during each visit to assess changes in subjective fullness ratings in response to perceived food availability. Higher scores indicate greater fullness.
Subjective satiety levels | On 1st and 2nd visit (after approximately 30 days)
  Subjective satiety levels are measured on a semi-continous scale from 1 (not at all) to 100 (extremely) repeatedly during each visit to assess changes in subjective satiety ratings in response to perceived food availability. Higher scores indicate greater satiation.
Subjective food cravings | On 1st and 2nd visit (after approximately 30 days)
  Subjective cravings for sweet, salty, and fatty foods are measured on a semi-continous scale from 1 (not at all) to 100 (extremely) repeatedly during each visit to assess changes in subjective food craving ratings in response to perceived food availability. Higher scores indicate stronger food craving.
Levels of diverse hormones | On 1st and 2nd visit (approximately 30 days later)
  Levels of different hormones (e.g., estradiol, progesteron, testosterone, ghrelin, leptin) will be measured via blood sampling.
Levels of cortisol | On 1st and 2nd visit (approximately 30 day later)
  Cortosol levels will be assessed multiple times throughout the visit as an objective measure of stress.
Insulin levels | On 1st and 2nd visit (after approximately 30 days)
  Levels of insulin will be measured multiple times throughout the visit via blood sampling.
Glucose levels | On 1st and 2nd visit (after approximately 30 days)
  Glucose levels will be measured multiple times throughout the visit via blood sampling.
Stress eating | On 1st and 2nd visit (after approximately 30 days)
  Changes in food intake related to stress is assessed with the Salzburg Stress Eating Scale (SSES; Meule et al., 2018). Higher Scores indicate increased food intake in response to stress, while lower scores indicate reduced food intake when experiencing stress.
Reward-related behavioral activation and inhibition | On 1st and 2nd visit (after approximately 30 days)
  Reward-related behavioral activation and inhibition are assessed using the Behavioral Inhibition System/Behavioral Activation System questionnaire (BIS/BAS; Strobel et al., 2001). Participants respond on a four-point Likert scale: "strongly disagree," "disagree," "agree," and "strongly agree." Higher scores on the BIS scale indicate greater behavioral inhibition, while higher scores on the BAS scale reflect stronger behavioral activation.
Impulsivity | On 1st and 2nd visit (after approximately 30 days)
  Impulsivity is assessed using the Barratt Impulsiveness Scale (BIS; Meule et al., 2011). Participants respond using a four-point scale: "rarely," "occasionally," "often," and "almost always." Higher scores indicate greater impulsivity.
Mood | On 1st and 2nd visit (after approximately 30 days)
  Mood is measured twice during each visit before and after the ad libitum meal using the Positive and Negative Affect Schedule (PANAS; Janke & Glöckner-Rist, 2014). Participants respond to 20 mood adjectives-10 reflecting positive affect and 10 reflecting negative affect-using a five-point scale: "not at all," "very slightly," "moderately," "quite a bit," and "extremely." Higher scores on the positive affect scale indicate stronger positive mood, while higher scores on the negative affect scale indicate stronger negative mood.
Emotion regulation | On 1st and 2nd visit (after approximately 30 days)
  Emotion regulation is assessed using the Emotion Regulation Questionnaire (ERQ; Abler & Kessler, 2009), which captures individual differences in the use of two distinct strategies to regulate emotions (cognitive reappraisal and expressive suppression). Participants rate their agreement with each item on a seven-point Likert scale, ranging from "strongly disagree" to "strongly agree." Higher scores on each subscale indicate more frequent use of the corresponding regulation strategy.
Perceived stress | On 1st and 2nd visit (after approximately 30 days)
  Perceived stress is assessed using the Perceived Stress Scale (PSS-10; Schneider et al., 2020), which aptures the extent to which individuals perceive their lives as unpredictable, uncontrollable, and overwhelming over the past month. Participants respond to general statements using a five-point scale ranging from "never" to "very often." Higher scores indicate greater perceived stress.
State anxiety | On 1st and 2nd visit (after approximately 30 days)
  State anxiety is assessed twice during each visit before and after the ad lib meal using the state version of the State-Trait Anxiety Inventory (STAI; Grimm, 2009); which captures the current intensity of anxiety as experienced at the moment of assessment. Response options include "almost never". "a little", "moderately", and "very much". Higher scores indicate higher levels of state anxiety.
Interoceptive awareness | On 1st and 2nd visit (after approximately 30 days)
  Interoceptive awareness is assessed using the Multidimensional Assessment of Interoceptive Awareness (MAIA; Eggart et al., 2021). The questionnaire measures various aspects of the awareness of internal bodily sensations. Participants respond to statements using a six-point scale: "never," "very rarely," "rarely," "occasionally," "frequently," and "always." Higher scores reflect greater awareness of bodily sensations.
Loss of control over eating | on 1st and 2nd visit (after approximately 30 days)
  Participants will rate their subjective loss of control over eating during the ad lib buffet task. Higher values indicate greater loss of control.

SECONDARY OUTCOMES:
Habitual food intake | On three days before the 1st visit
  Self-reported habitual food intake (i.e., all food and drinks consumed) is assessed via an app and/or through additional handwritten food diaries on three consecutive days.
Quantification of epigenetic markers related to appetite, menstrual cycle, and stress | On 1st and 2nd visit (after approximately 30 days)
  Epigenetic markers associated with appetite regulation, menstrual function, and stress response will be measured in blood samples. Site-specific epigenetic modifications (e.g., DNA methylation or histone modifications) will be quantified using validated molecular assays.
Depressive mood | On 1st and 2nd visit (after approximately 30 days)
  Depressive mood is assessed using the German version of the Beck Depression Inventory (BDI; Kühner et al., 2007). The questionnaire measures the severity of depressive symptoms experienced over the past two weeks. Higher total scores indicate more pronounced depressive symptomatology.
Body image | On 1st and 2nd visit (after approximately 30 days)
  Body image is assessed using the Body Shape Questionnaire (BSQ; Pook et al., 2008), which measures concerns related to body shape commonly associated with eating disorders. Participants rate how frequently they experience body-related thoughts and feelings. Higher scores indicate greater body shape concern.
Trait food cravings | On 1st and 2nd visit (after approximately 30 days)
  Food cravings are measured using the trait version of the Food Cravings Questionnaire (FCQ-T; Meule et al., 2012). Responses are given on a six-point scale from "never/not applicable" to "always," with higher scores indicating more frequent and intense cravings.
Dietary patterns | Day 2 (after approximately 30 days after day 1 i.e., 1st visit)
  Dietary patterns are assessed using a food frequency questionnaire (Haftenberger et al., 2018), which captures the frequency and quantity of consumption across various foods and food groups over the past month. Participants indicate how often they consumed specific items and in which quantity, allowing for an overview of habitual dietary intake and eating patterns.
Intuitive eating | On 1st and 2nd visit (after approximately 30 days)
  Intuitive eating is assessed using the Intuitive Eating Scale-2 (van Dyck et al., 2019), which evaluates individuals' tendency to rely on physical hunger and satiety cues to guide decisions about when, what, and how much to eat. Participants respond on a five-point scale ranging from "strongly disagree" to "strongly agree." Higher scores reflect a greater inclination toward intuitive eating behaviors.
Food insecurity status | On 1st and 2nd visit (after approximately 30 days)
  Food insecurity status is assessed using the Food Insecurity Experience Scale (FIES; Depa et al., 2018), which evaluates individuals' access to food by addressing factors such as financial constraints, availability, and dietary quality. Response options include "yes," "no," "refused," and "don't know." Higher scores reflect greater severity of food insecurity.
Restrained eating | Day 1 (1st visit out of 2)
  Restrained eating is assessed using the "Cognitive Restraint of Eating" subscale from the Three-Factor Eating Questionnaire (TFEQ; Pudel & Westenhöfer, 1989). The subscale includes both true/false items and statements rated on a four-point Likert scale ranging from 1 ("always") to 4 ("never"). Higher total scores indicate greater cognitive restraint in eating behavior.
Eating motives | Day 1 (1st visit out of 2)
  Eating motives will be assessed using the Eating Motives Survey (TEMS; Renner et al., 2012). Items are rated on a 7-point Likert scale, ranging from "never" to "always". Higher scores on TEMS subscales indicate a greater reliance on those eating motives when making food or eating choices.
Family climate | Day 1 (1st visit out of 2)
  Family climate is measured using the Familien Klima Skale (FKS; Roth, 2003). Items are rated on a 5-point Likert scale ranging from 1) "does not apply at all," 2) "applies little," 3) "applies moderately," 4) "applies predominantly," to 5) "applies almost completely." Higher total scores indicate a better family climate.
Attachment styles | Day 1 (1st visit out of 2)
  Attachment styles will be assessed using the Adult Attachment Scale (AAS; Schmidt et al., 2004). Items are rated on a five-point Likert scale ranging from "not at all true" to "exactly true." Higher scores on each subscale indicate a stronger endorsement of the corresponding attachment dimension. The subscales/attachment styles assessed are secure, avidant, anxious.
Gut Microbiome | 1 to three days before the 1st visit
  To assess the relationship between the gut microbiome and participants' food intake during the ad libitum meal, fecal samples will be collected prior to the first visit, during the observational phase in which participants record their habitual dietary intake.

CONTACTS AND LOCATIONS:
Overall Officials: Soyoung Q Park, Prof. Dr., Principal Investigator — German Institute of Human Nutrition Potsdam-Rehbruecke
Locations (1):
- German Institute of Human Nutrition Potsdam-Rehbruecke, Nuthetal, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haftenberger M, Heuer T, Heidemann C, Kube F, Krems C, Mensink GB. Relative validation of a food frequency questionnaire for national health and nutrition monitoring. Nutr J. 2010 Sep 14;9:36. doi: 10.1186/1475-2891-9-36. PMID 20840739
- [Background] Langenbach BP, Baumgartner T, Cazzoli D, Muri RM, Knoch D. Inhibition of the right dlPFC by theta burst stimulation does not alter sustainable decision-making. Sci Rep. 2019 Sep 25;9(1):13852. doi: 10.1038/s41598-019-50322-w. PMID 31554883
- [Background] Teslovich T, Freidl EK, Kostro K, Weigel J, Davidow JY, Riddle MC, Helion C, Dreyfuss M, Rosenbaum M, Walsh BT, Casey BJ, Mayer L. Probing behavioral responses to food: development of a food-specific go/no-go task. Psychiatry Res. 2014 Sep 30;219(1):166-70. doi: 10.1016/j.psychres.2014.04.053. Epub 2014 May 10. PMID 24909971
- [Background] Schmidt S, Strauss B, Hoger D, Brahler E. [The Adult Attachment Scale (AAS) - psychometric evaluation and normation of the German version]. Psychother Psychosom Med Psychol. 2004 Sep-Oct;54(9-10):375-82. doi: 10.1055/s-2003-815000. German. PMID 15343479
- [Background] Renner B, Sproesser G, Strohbach S, Schupp HT. Why we eat what we eat. The Eating Motivation Survey (TEMS). Appetite. 2012 Aug;59(1):117-28. doi: 10.1016/j.appet.2012.04.004. Epub 2012 Apr 19. PMID 22521515
- [Background] Depa J, Gyngell F, Muller A, Eleraky L, Hilzendegen C, Stroebele-Benschop N. Prevalence of food insecurity among food bank users in Germany and its association with population characteristics. Prev Med Rep. 2018 Jan 28;9:96-101. doi: 10.1016/j.pmedr.2018.01.005. eCollection 2018 Mar. PMID 29527460
- [Background] Meule A, Lutz A, Vogele C, Kubler A. Food cravings discriminate differentially between successful and unsuccessful dieters and non-dieters. Validation of the Food Cravings Questionnaires in German. Appetite. 2012 Feb;58(1):88-97. doi: 10.1016/j.appet.2011.09.010. Epub 2011 Sep 29. PMID 21983051
- [Background] Pook M, Tuschen-Caffier B, Brahler E. Evaluation and comparison of different versions of the Body Shape Questionnaire. Psychiatry Res. 2008 Feb 28;158(1):67-73. doi: 10.1016/j.psychres.2006.08.002. Epub 2007 Nov 26. PMID 18037499
- [Background] Kuhner C, Burger C, Keller F, Hautzinger M. [Reliability and validity of the Revised Beck Depression Inventory (BDI-II). Results from German samples]. Nervenarzt. 2007 Jun;78(6):651-6. doi: 10.1007/s00115-006-2098-7. German. PMID 16832698
- [Background] Eggart M, Todd J, Valdes-Stauber J. Validation of the Multidimensional Assessment of Interoceptive Awareness (MAIA-2) questionnaire in hospitalized patients with major depressive disorder. PLoS One. 2021 Jun 25;16(6):e0253913. doi: 10.1371/journal.pone.0253913. eCollection 2021. PMID 34170963
- [Background] Schneider EE, Schonfelder S, Domke-Wolf M, Wessa M. Measuring stress in clinical and nonclinical subjects using a German adaptation of the Perceived Stress Scale. Int J Clin Health Psychol. 2020 May-Aug;20(2):173-181. doi: 10.1016/j.ijchp.2020.03.004. Epub 2020 May 22. PMID 32550857
- [Background] Meule A, Reichenberger J, Blechert J. Development and preliminary validation of the Salzburg Stress Eating Scale. Appetite. 2018 Jan 1;120:442-448. doi: 10.1016/j.appet.2017.10.003. Epub 2017 Oct 3. PMID 28986162
- [Background] Gueguen MCM, Anllo H, Bonagura D, Kong J, Hafezi S, Palminteri S, Konova AB. Recent Opioid Use Impedes Range Adaptation in Reinforcement Learning in Human Addiction. Biol Psychiatry. 2024 May 15;95(10):974-984. doi: 10.1016/j.biopsych.2023.12.005. Epub 2023 Dec 13. PMID 38101503
- [Background] Liu L, Artigas SO, Ulrich A, Tardu J, Mohr PNC, Wilms B, Koletzko B, Schmid SM, Park SQ. Eating to dare - Nutrition impacts human risky decision and related brain function. Neuroimage. 2021 Jun;233:117951. doi: 10.1016/j.neuroimage.2021.117951. Epub 2021 Mar 12. PMID 33722669
- [Background] Eisenstein SA, Gredysa DM, Antenor-Dorsey JA, Green L, Arbelaez AM, Koller JM, Black KJ, Perlmutter JS, Moerlein SM, Hershey T. Insulin, Central Dopamine D2 Receptors, and Monetary Reward Discounting in Obesity. PLoS One. 2015 Jul 20;10(7):e0133621. doi: 10.1371/journal.pone.0133621. eCollection 2015. PMID 26192187
- See also: Abler, B. & Kessler, H. (2011). ERQ. Emotion Regulation Questionnaire [Verfahrensdokumentation aus PSYNDEX Tests-Nr. 9006192 und Fragebogen]. In Leibniz-Zentrum für Psychologische Information und Dokumentation (ZPID) (Hrsg.), Elektronisches Testarchiv. — https://doi.org/10.23668/psycharchives.6497
- See also: Janke, S., & Glöckner-Rist, A. (2012). Deutsche Version der Positive and Negative Affect Schedule (PANAS). Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS). — https://doi.org/10.6102/zis146
- See also: Grimm, Jürgen (Hg.) (2009): State-Trait-Anxiety Inventory nach Spielberger. Deutsche Lang- und Kurzversion.- Methodenforum der Universität Wien. MF-Working Paper 2009/02 — https://empcom.univie.ac.at/fileadmin/user_upload/p_empcom/pdfs/Grimm2009_StateTraitAngst_MFWorkPaper2009-02.pdf
- See also: Van Dyck, Z., Herbert, B. M., Happ, C., Kleveman, G. V., & Vögele, C. (2019). IES-2. Deutsche Version der Intuitive Eating Scale 2 [Verfahrensdokumentation und Fragebogen]. In Leibniz-Institut für Psychologie (ZPID) (Hrsg.), Open Test Archive. Trier: ZPI — https://doi.org/10.23668/psycharchives.15697
- See also: Pudel V., Westenhöfer, J. (1989): Fragebogen zum Essverhalten. F-E-V, Hogrefe, Göttingen. — https://www.testzentrale.de/shop/fragebogen-zum-essverhalten.html
- See also: Roth, M.(2003). Kurzform der Familienklimaskalen für Jugendliche. Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS). — https://doi.org/10.6102/zis195